CLINICAL TRIAL: NCT03223727
Title: Registry of Treatment Outcomes in a Non-study Population of Symptomatic Metastasized Castration Resistant Prostate Cancer (mCRPC) Patients Treated With Radium-223
Brief Title: Treatment Outcomes in a Non-study Population of Symptomatic mCRPC Patients Treated With Radium-223
Acronym: ROTOR
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: m15RTO
Record Dates: First submitted 2017-04-04; First posted 2017-07-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer Metastatic; Bone Metastases
Keywords: Radium-223
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Extra blood will be collected at baseline, 1st, 2nd, 3rd and 6th (or last) Radium-223 treatment. Changes in serum and blood levels of biomarkers of bone metabolism and levels of blood osteoclast precursors in Radium-223 treated patients will e evaluated for their potential to predict treatment outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood tests — Blood tests for several bone markers (see summary)

SUMMARY:
This registry aims to evaluate the efficacy of Rad-223 treatment in a non-study population of CRPC patients treated earlier with Docetaxel and patients not treated earlier with Docetaxel and efficacy of the first subsequent therapy. The indication for treatment with Radium-223 will be at the physician's decision. All patients treated with Radium-223 can be included in this registry. The registry only dictates the collection of base line characteristics, expansion of regular blood tests and patient reported pain scores.

DETAILED DESCRIPTION:
Serum and blood markers of bone metabolism will be evaluated at Base Line, 1st, 2nd, 3rd and 6th (or last) Radium- 223 treatment. Every blood draw prior to Radium-223 treatment At baseline, tests include (but not restricted to): Testosterone, vitamin D-25-OH (Calciferol), C-reactive protein, Rank Ligand, IL6, BSAF, P1NP and CTX. Patients need to be fasting when blood is collected. (2x8,5 ml gel tube; Limited to 100 patients in selected centres). Before 2nd, 3rd, 4th and 6th (or last) Radium-223 treatment, tests include (but not restricted to): C-reactive protein, Rank, Ligand, IL6, BSAF, P1NP and CTX. Patients need to be fasting when blood is collected. (2x8,5 ml gel tube; Limited to 100 patients in selected centers).

Moreover, levels of osteoclast precursors (CD34+) will be evaluated (10 ml heparinized blood) prior to the first Radium-223 treatment, 3rd and last treatment (Limited to 100 patients in selected centres).

All above-mentioned blood collections will be from the same venipuncture as standard clinical labs. Experimental assessments will be evaluated for their value as biomarkers of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* At the physicians discretion
* Age 18 year and older.
* Written informed consent

Exclusion Criteria:

* Previous treatment with Radium-223.
* Participation in another Radium-223 study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer and bone metastasis, which are to be treated with Radium-223.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment on pain outcomes, as mentioned by the patient | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate Radium-223 treatment efficacy by patient, by several questionnaires (FACT-P, BPI-S and use of painmedication).
Efficacy of treatment by patient records | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  But also by patient records (records of bonescans, CT scans, blood measurements, out-patient clinic visits).
  All of these assessments will be combined to come to a final reported value (Progressive disease, stable disease, partial remission or complete remission)

SECONDARY OUTCOMES:
Symptomatic Skeletal Event | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  To evaluate the efficacy of Radium-223 treatment in a nonstudy population by effects on Symptomatic Skeletal Event (SSE). Through patient records and questionnairs (FACT-P, BPI-S and use of painmedication).
Clinical Parameters assessed by the WHO PS. | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate Radium-223 treatment efficacy in a non-study population of CRPC patients by clinical parameters, through patient records (WHO PS)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate Radium-223 treatment tolerability in a non-study population of CRPC patients, through patient records (using the CTCAE v4.03 for adverse events).
Subsequent therapy after Radium-223: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate of the treatment after Radium-223 the treatment tolerability in a non-study population of CRPC patients, through patient records (using the CTCAE v4.03 for adverse events).
Biomarkers | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Identification of predictive clinical and explorative biomarkers of Radium-223 efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Andre Bergman, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- Netherlands (2):
  - The Netherlands Cancer Intitute, Amsterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam